CLINICAL TRIAL: NCT02099006
Title: Novel Topical Therapies for the Treatment of Genital Pain
Acronym: Topicals
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Mae Stone Goode Foundation (Other)
Responsible Party: Principal Investigator, Adrienne Bonham, Associate Professor, University of Rochester
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 46905
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Results first posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Female Genital Diseases
MeSH Terms: conditions — Genital Diseases, Female | interventions — Amitriptyline; Baclofen; Ketoprofen; Ketamine; Loperamide; bismuth subsalicylate; Gabapentin; cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medications (Experimental): Each study subject will be sequentially exposed to each of the study drugs and the placebo in a random order. The study is designed as a double blinded, crossover study.
  Interventions: Drug: Amitriptyline; Drug: Baclofen; Drug: Ketoprofen; Drug: Ketamine; Drug: Loperamide; Drug: Gabapentin
- Placebo (Placebo Comparator): The compounding base alone will be used as a placebo. Each participant will be given each drug and the placebo sequentially in random order.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Amitriptyline — Topical application of the drug at a 2% concentration in combination with 2% Baclofen
  Other Names: Elavil
  Arms: Medications
Drug: Baclofen — Used topically at 2% concentration in combination with 2% amitriptyline
  Other Names: Lioresal
  Arms: Medications
Drug: Ketoprofen — To be applied topically at a 10% concentration
  Other Names: Orudis; Oruvail; Nexcede; Orudis KT
  Arms: Medications
Drug: Ketamine — To be applied topically at a 10% concentration
  Other Names: Ketalar
  Arms: Medications
Drug: Loperamide — To be applied topically at a 5% concentration
  Other Names: Imodium; Imotil; Kaopectate
  Arms: Medications
Drug: Gabapentin — To be applied topically at a 6% concentration
  Other Names: Neurontin
  Arms: Medications
Drug: placebo — Compounding base to be used alone as a placebo
  Other Names: Cetaphil
  Arms: Placebo

SUMMARY:
This study is testing drugs not previously used topically for the treatment of vulvodynia, a common genital pain syndrome. It is hoped that one of these drugs will improve vaginal entryway pain with touch, daily pain scores and sexual functioning.

DETAILED DESCRIPTION:
Vulvodynia is defined as burning pain, occurring in the absence of any visible finding or a clinically identifiable nervous disorder. Current treatments include vulvar care measure, topical medications, oral medications, biofeedback, physical therapy and surgery. The usual treatment is to have the patient take either tricyclic antidepressants or anti convulsants orally, however these methods seldom bring total relief. These drugs do have significant side effects limiting the patient's tolerance of the higher does sometimes needed. An effective topical medication would greatly benefit these women with fewer side effects and better tolerance. Topical amitriptyline and baclofen are often prescribed, but no studies have been done to support their use. Topical gabapentin has also been shown to have good effect, but no prospective clinical study as been done.

This study will test topical application of Cetaphil, Loperamide, Gabapentin, Ketoprofen, Ketamine and Amitriptyline over a 19 week period in the first phase of the study. The drugs are compounded by the University of Rochester research pharmacy and dispensed in 19 vials, one vial to be used each week. Patients and study personnel are blinded as to which drug is being used. Each study participant was given a week of placebo at the initiation of the study. Each study compound, which contains both the drug and the base (Cetaphil) will be used twice a day for two weeks in a row, followed by a one week washout of base alone. If a patient finds that one of the drugs is effective she may stop participation after the first 13 weeks and request that the most effective drug be prescribed for her. The unblinding officer would then work with the research pharmacy to identify the effective drug and provide the patient with a prescription for that drug. If the patient desires, she may enroll in the second phase of the study when she will test the last two drugs over a six week period with the washout as in the first segment of the study. The drugs would be administered in vials as in the first section of the study.

Every week on Sunday the patient will complete an electronic diary, recording her daily pain, any drug side effects, pain with the tampon test and overall health. Every three weeks she will complete the Female Sexual Function Index on the same electronic system. She would start her new drug on Monday each week. Additionally the coordinator of the study will call each patient on Wednesday to see if they are having any problems with the drug started on Monday.

All patients who could become pregnant are required to maintain effective contraception throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Women between ages of 18 and 65 who complain of localized provoked vulvar pain and meet the criteria for the diagnosis of localized provoked vulvodynia. Patients who have failed or have been unable to tolerate previous attempts at systematic therapy or surgery will be specifically recruited.

Exclusion Criteria:

1. The presence of a dermatologic or neurologic condition which is determined by the investigator to be the primary cause of the patient's pain.
2. Allergy to any of the medications or the base itself.
3. Concurrent use of the following medications. . The patient may enroll in the study after a two week washout from these medications. Patients may need to receive approval from the prescribing physician before stopping these medications. Failure to obtain approval for medication cessation would be cause for exclusion.

Gabapentin (NeurontinTM) Amitriptyline (ElavilTM) Nortriptyline (PamelorTM) Desipramine (NorpraminTM) Tramadol (UltramTM, ConZipTM, RybixTM, RysoltTM, Ultram ERTM) Pregabalin (LyricaTM) Baclofen

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne D Bonham, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Each study subject was sequentially exposed to each of the study drugs and the placebo in a random order. The study is designed as a double blinded, crossover study.
  Amitriptyline 2%/ Baclofen 2%: Topical application of the drug at a 2% concentration in combination with 2% Baclofen
  Ketoprofen: To be applied topically at a 10% concentration
  Ketamine: To be applied topically at a 10% concentration
  Loperamide: To be applied topically at a 5% concentration
  Gabapentin: To be applied topically at a 6% concentration
Period: Overall Study
Arm/Group | All Study Participants
Started | 9
Received Placebo | 9
Received Amitriptyline/ Baclofen | 7
Received Ketoprofen | 3
Received Loperamide | 7
Received Ketamine | 6
Received Gabapentin | 8
Completed | 8
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Each study subject will be sequentially exposed to each of the study drugs and the placebo in a random order. The study is designed as a double blinded, crossover study.
  Amitriptyline/ Baclofen: Topical application of the drug at a 2% concentration in combination with 2% Baclofen
  Ketoprofen: To be applied topically at a 10% concentration
  Ketamine: To be applied topically at a 10% concentration
  Loperamide: To be applied topically at a 5% concentration
  Gabapentin: To be applied topically at a 6% concentration
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Daily Genital Pain.
Description: Each subject was asked to keep a symptom diary recording her daily genital pain, measured on a 10 point Likert scale. A score of "0" was defined as no pain and a score of "10" was defined as worst imaginable pain. These daily values were collected and a mean pain score for the period of treatment was calculated.
Time Frame: 13 weeks
Population: For each placebo entry the data is limited to include only those participates who also received the named intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medications | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale
  Loperamide | 2.4 (1.94) | 2.92 (2.3)
  Ketamine | 3.42 (2.45) | 2.77 (2.46)
  Gabapentin | 3.70 (2.92) | 3.41 (2.55)
  amtriptyline/baclofen | 3.87 (2.74) | 3.61 (2.68)
  ketoprofen | 5.05 (3.34) | 5.05 (3.45)
Statistical Analysis 1: Comparison: Medications vs Placebo; Null hypothesis - that the improvement in daily genital pain would be no different with the daily application of loperamide than with the daily application of a placebo cream; Test type: Superiority or Other; p = 0.30, t-test, 2 sided; Paired T test
Statistical Analysis 2: Comparison: Medications vs Placebo; Null hypothesis - that the improvement in daily genital pain would be no different with the daily application of ketamine than with the daily application of a placebo cream; Test type: Superiority or Other; p = 0.33, t-test, 2 sided; Paired
Statistical Analysis 3: Comparison: Medications vs Placebo; Null hypothesis - that the improvement in daily genital pain would be no different with the daily application of gabapentin than with the daily application of a placebo cream; Test type: Superiority or Other; p = 0.65, t-test, 2 sided; paired
Statistical Analysis 4: Comparison: Medications vs Placebo; Null hypothesis - that the improvement in daily genital pain would be no different with the daily application of amitriptyline and baclofen than with the daily application of a placebo cream; Test type: Superiority or Other; p = 0.25, t-test, 2 sided; Paired
Statistical Analysis 5: Comparison: Medications vs Placebo; Null hypothesis - that the improvement in daily genital pain would be no different with the daily application of ketoprofen than with the daily application of a placebo cream; Test type: Superiority or Other; p = 1.0, t-test, 2 sided; Paired

2. Secondary Outcome: Reduction in Tampon Test Pain
Description: Reduction in the pain, as measured on a 10 point Likert scale, associated with the insertion and removal of a tampon. This is a validated surrogate for pain associated with intercourse. Subjects were asked to insert and remove a tampon each week and report the degree of pain associated with this. A score of "0" was defined as no pain, and a score of "10" was defined as worst imaginable pain.
Time Frame: 13 weeks
Population: For each placebo entry the data is limited to include only those participates who also received the named intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medications | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale
  loperamide | 4.71 (2.75) | 5.29 (3.21)
  ketamine | 5.92 (3.56) | 5.92 (3.00)
  gabapentin | 5.125 (3.57) | 4.875 (3.19)
  ketoprofen | 6.17 (3.18) | 6.0 (3.46)
  amitriptyline/baclofen | 5.43 (2.75) | 5.36 (3.12)
Statistical Analysis 1: Comparison: Medications vs Placebo; Null hypothesis - that the improvement in tampon test pain would be no different with the daily application of loperamide cream than with the daily application of a placebo cream; Test type: Superiority or Other; p = 0.31, t-test, 2 sided; paired
Statistical Analysis 2: Comparison: Medications vs Placebo; Null hypothesis - that the improvement in tampon test pain would be no different with the daily application of ketamine cream than with the daily application of a placebo cream; Test type: Superiority or Other; p = 1, t-test, 2 sided; Paired
Statistical Analysis 3: Comparison: Medications vs Placebo; Null hypothesis - that the improvement in tampon test pain would be no different with the daily application of gabapentin cream than with the daily application of a placebo cream; Test type: Superiority or Other; p = 0.66, t-test, 2 sided; Paired
Statistical Analysis 4: Comparison: Medications vs Placebo; Null hypothesis - that the improvement in tampon test pain would be no different with the daily application of ketoprofen cream than with the daily application of a placebo cream; Test type: Superiority or Other; p = 0.42, t-test, 2 sided; Paired
Statistical Analysis 5: Comparison: Medications vs Placebo; Null hypothesis - that the improvement in tampon test pain would be no different with the daily application of amitriptyline/baclofen cream than with the daily application of a placebo cream; Test type: Superiority or Other; p = 0.79, t-test, 2 sided; Paired

ADVERSE EVENTS:
Time Frame: 1.5 years
Arm/Group | Medications | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
The small number of patients recruited left this study underpowered to uncover significant effects with the medications studied.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes